CLINICAL TRIAL: NCT05831917
Title: MRI - Guided Adaptive RadioTHerapy for Dysphagia in Head and Neck Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sichuan Cancer Hospital and Research Institute (Other)
Responsible Party: Principal Investigator, Yangkun Luo, Study Director, Sichuan Cancer Hospital and Research Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SCCHEC-02-2023-017
Record Dates: First submitted 2023-04-16; First posted 2023-04-26 (Actual); Last update posted 2023-04-26 (Actual); Status verified 2023-04

CONDITIONS: HNSCC
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck | interventions — Radiotherapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment Group (Experimental)
  Interventions: Radiation: Radiotherapy

INTERVENTIONS:
Radiation: Radiotherapy — Radiotherapy: All patients were treated with Unity MRI Linac intensity modulated radiation therapy, daily imaging of MRI-IGRT and online target delineation, redesign, and total radiation dose: GTV 70Gy/33f, GTVLN 70Gy/33f, CTV 60Gy/33f, CTVLN 54Gy/33f, 5 days per week. Dose limit: The average dose to the upper, middle, and lower pharyngeal constrictor muscles is ≤ 40-50Gy, with oropharyngeal cancer requiring an average dose to the upper, middle, and lower pharyngeal constrictor muscles to be ≤ 50Gy and ≤ 20Gy; Lower pharyngeal cancer requires an average dose of ≤ 40Gy for the upper and middle pharyngeal constrictor muscles, and ≤ 50Gy for the lower pharyngeal constrictor muscles.
  chemotherapy: cisplatin 75mg/m2, 21 days per cycle, a total of 3 cycles.

SUMMARY:
Recently developed hybrid machines (MRidian®-CE approval since 2016), consisting of a linear accelerator and an integrated low-field MRI, could allow better visualization of tumor and organs at risk during patient positioning and daily treatment finally repetitive adaptation of target volumes according to changes in patient weight and tumor anatomy during the radiotherapy course. These procedures would facilitate a high-precision treatment and help reduce dose exposure of critical structures.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-70 years old;
2. I-IVb stage oral cancer, hypopharyngeal cancer, laryngeal cancer, oropharyngeal cancer confirmed by histopathology or cytology (AJCC 8th edition);
3. Receiving radical synchronous radiotherapy and chemotherapy;
4. According to the RECIST version 1.1 evaluation criteria, at least one measurable lesion is present;
5. ECOG PS score 0-1;
6. Hematology indicators are basically normal: white blood cell count ≥ 4 × 109/L； Absolute neutrophil count ≥ 1.5 × 109/L； Platelets ≥ 100 × 109/L； Hemoglobin ≥ 90g/L; Kidney function is basically normal: serum creatinine ≤ 1.5 × ULN or creatinine clearance rate (CrCl)>60 mL/min (using Cockcroft Fault formula): Female CrCl=(140 age) × Body weight (kg) × 0.85 / (72 × Scr mg/dl)； Male CrCl=(140 age) × Body weight (kg) × 1.00 / (72 × Scr mg/dl) Liver function is basically normal: serum total bilirubin ≤ 1.5 × ULN； Cereal grass transaminase (AST) ≤ 2.5 × ULN； Glutamate transaminase (ALT) ≤ 2.5 × ULN；
7. Having sufficient cognitive ability to complete the questionnaire survey;
8. Able to understand and willing to sign a written informed consent form.

Exclusion Criteria:

1. There is evidence of swallowing dysfunction (unrelated to HNSCC);
2. Patients who have previously received radiotherapy for the head and neck region;
3. Recurrent or metastatic patients;
4. Involvement of posterior pharyngeal wall, posterior ring, and posterior pharyngeal lymph nodes;
5. Previous tumor resection surgery or major head and neck surgery (excluding biopsy/tonsillectomy);
6. Previous tracheotomy;
7. Participated in other interventional clinical trials within 30 days prior to screening;
8. Individuals with a history of other malignant tumors (excluding cured skin basal cell carcinoma)
9. There are concurrent diseases with poor control (such as heart failure, severe lung disease, severe liver disease, mental illness, etc.);
10. Individuals who are allergic to the use of drugs or their components in this protocol;
11. Pregnant (confirmed by blood or urine HCG testing) or lactating women, or subjects of childbearing age who are unwilling or unable to take effective contraceptive measures (applicable to both male and female subjects) until at least 6 months after the last trial treatment;
12. Researchers believe that it is not suitable to participate in this study;
13. Those who are unwilling to participate in this study or unable to sign an informed consent form;

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Estimated)
Dates: Start 2023-01-17 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
Swallowing Difficulty | 12 months
  Swallowing Difficulty will be assessed by MDADI swallowing difficulty score

CONTACTS AND LOCATIONS:
Locations (1):
- Sichuan Cancer Hospital and Research Institute, Chengdu, Sichuan, China